CLINICAL TRIAL: NCT00100438
Title: Incidence of Parkinson's Disease Among Veterans
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: Epid-013-98S
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
This is a database study. Medical records will be reviewed in order to document a new or pending diagnosis of Parkinson's disease and in order to learn more about the disease process. Other than the time that it takes to complete a medical record authorization form, no other human subject participation will be needed.

ELIGIBILITY:
chart review

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs Medical Center, Houston, Texas, United States